CLINICAL TRIAL: NCT04838782
Title: Role of Repeat Resection in Recurrent Glioblastoma (4rGBM) Trial: a Randomized Care Trial for Patients With Recurrent GBM
Brief Title: Role of Repeat Resection in Recurrent Glioblastoma
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient patient population
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CC-210049
Record Dates: First submitted 2021-04-04; First posted 2021-04-09 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Recurrent Glioblastoma; Glioblastoma - Category
Keywords: rGBM, repeat GBM, recurrent high grade astrocytoma
MeSH Terms: conditions — Glioblastoma; Astrocytoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Repeat Surgical Resection (Experimental): Standard surgical operative management according to local practices.
  Interventions: Procedure: Repeat Surgical Management of Recurrent GBM
- Management Without Re-operation (Active Comparator): Non-surgical management with standard care according to local practices.
  Interventions: Procedure: Repeat Surgical Management of Recurrent GBM

INTERVENTIONS:
Procedure: Repeat Surgical Management of Recurrent GBM — Routine of surgical operative management. Details of treatment will be left to local centers, and recorded in the case report form (CRF).

SUMMARY:
Patients with recurrent Glioblastoma (GBM) are commonly presented to surgeons, along with the question of whether or not to re-resect the recurrence. There is no Level 1 evidence to support a role for repeat surgery in this context, but a multitude of observational research suggests that repeat surgery may improve quality survival. Unfortunately, these studies all suffer from selection bias.

The goal of this study is to provide a care trial context to help neurosurgeons manage patients presenting with recurrent GBM, with no additional risks, tests, or interventions than what they would normally encounter in routine care. Secondary goals include a test of the hypothesis that repeat resection can improve median overall survival, and that it can increase the number of days of survival outside of a hospital/nursing/palliative care facility.

DETAILED DESCRIPTION:
Glioblastoma (GBM) is the most common malignant brain tumor (48.3% of malignant tumors).1 It has a predilection for Caucasian men with a mean age of 65.1, 2 There are approximately 13,000 new diagnoses of GBM made every year in the United States.1 Patients have an average survival of 12-15 months, with a 5-year survival rate of 6.8% despite various treatments.1 If the prognosis at the time of initial diagnosis is grim, it is even worse at the time of recurrence. Recurrence after the initial resection, which can be symptomatic or discovered on surveillance MRI imaging, occurs in nearly all patients, usually within the first year, even when the initial management is aggressive.3-6 There is no standard way to care for recurrent GBM patients and treatment may include one or more of the following: repeat surgery, radiation therapy, or second-line chemotherapy.7

Repeat surgical management carries a greater risk of wound infection and cerebrospinal fluid leak than the initial surgery, especially in patients who received radiation.8 When maximal resection was attempted at the time of the initial procedure, the second surgery is more at risk of neurological injury. Repeat surgical management often also entails a delay in the initiation of further chemotherapy, as these agents are not administered peri-operatively because of potentially deleterious effects on wound healing. Nonetheless, despite, or because of the desperate setting, patients and surgeons are often pressed to consider repeat surgery, which is performed in at least 10-30% of patients.9 Repeat surgical treatment may be more favorable with younger age (<60 years), and preoperative Karnofsky performance status (KPS) of at least 70.9 Median survival following repeat resection varies between 13-54 weeks,10, 11 but all reports suffer from the limitations of retrospective studies, the most obvious being selection bias in terms of patient age, functional status, tumor location and size.11, 12 Yet, despite favorable biases some studies report no improvement in terms of survival or quality of life.13, 14 Two recent systematic meta-analyses of case series offer conflicting conclusions about the merit of re-operation.15, 16

If the intent of repeat surgery is to improve quality and quantity of life, there is no level 1 evidence it is effective.3, 16, 17 Thus repeat surgery should be considered the experimental arm of a randomized trial designed in the best interest of the patient, being only offered as a 50% chance, always balanced by a 50% chance of being allocated non-surgical care, or a chance to escape what could turn out to be unnecessary or harmful surgery.18 For patients may be better served by being free to pursue other life priorities in the company of loved ones rather than being scheduled to endure repeat craniotomy and multiple clinical or research follow-up visits. There is sufficient community equipoise to support the conduct of such a randomized trial.19

Tria Design:

The trial is a simple, all-inclusive, prospective, multicenter, randomized care trial18 that allocates 1:1 re-operation (or not) for patients with recurrent Glioblastoma. The primary outcome is overall survival. Secondary outcomes include standard peri-operative safety outcomes and (a notion of) 'quality survival', or survival at home, measured by counting days of survival minus days in hospital/nursing home/palliative care setting. Blinding is not feasible; treatment allocation will not be masked. The trial allows for pre-randomization.22 The burden of the proof of benefit is on surgery. While some patients allocated non-surgical management may still want surgery, and some patients allocated surgery may prefer non-surgical management, we feel participating patients will be better informed by the discussion around trial participation.

Hypothesis:

Patients with recurrent Glioblastoma, at the time they are considered for repeat resection, who undergo repeat resection for the GBM, will experience an increase in median overall survival from 6 to 9 months.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Previously histologically confirmed and surgically resected Glioblastoma
* Previous craniotomy for open tumor resection (needle biopsies alone do not count as resection)
* The attending surgeon considers re-operation may improve quality survival

Exclusion Criteria:

* Informed consent not possible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-08-26 (Actual); Primary Completion 2025-03-24 (Actual); Study Completion 2025-03-24 (Actual)

PRIMARY OUTCOMES:
Length of Overall Survival | Follow-up for 5 Years or until death
  The primary outcome is time to death from any cause, starting from the time of inclusion.

SECONDARY OUTCOMES:
Total length of hospitalization / palliative care / nursing home | Follow-up for 5 Years or until death
Discharge to a location other than home | Follow-up for 5 Years or until death
Total number of days spent outside a hospital or nursing care facility. | Follow-up for 5 Years or until death
Incidence of peri-operative non-neurological complications (wound infection, CSF leaks) | Follow-up for 5 Years or until death
Incidence of new significant neurological deficits after surgery (defined as new or substantially worsened aphasia, or new weakness (MRC power < 3 in one or more limbs). | Follow-up for 5 Years or until death

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta Division of Neurosurgery, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available upon reasonable request.
Supporting Information: Study Protocol, ICF
Time Frame: Indefinitely

REFERENCES:
- [Background] Ostrom QT, Cioffi G, Gittleman H, Patil N, Waite K, Kruchko C, Barnholtz-Sloan JS. CBTRUS Statistical Report: Primary Brain and Other Central Nervous System Tumors Diagnosed in the United States in 2012-2016. Neuro Oncol. 2019 Nov 1;21(Suppl 5):v1-v100. doi: 10.1093/neuonc/noz150. PMID 31675094
- [Background] Thakkar JP, Dolecek TA, Horbinski C, Ostrom QT, Lightner DD, Barnholtz-Sloan JS, Villano JL. Epidemiologic and molecular prognostic review of glioblastoma. Cancer Epidemiol Biomarkers Prev. 2014 Oct;23(10):1985-96. doi: 10.1158/1055-9965.EPI-14-0275. Epub 2014 Jul 22. PMID 25053711
- [Background] Yahia-Cherif, M., De Witte, O., Mélot, C., & Lefranc, F. (2019). P14.56 Recurrent Glioblastomas: Should we operate a second and even a third time. Neuro-Oncology, 21(Suppl 3), iii80.
- [Background] De Bonis P, Anile C, Pompucci A, Fiorentino A, Balducci M, Chiesa S, Lauriola L, Maira G, Mangiola A. The influence of surgery on recurrence pattern of glioblastoma. Clin Neurol Neurosurg. 2013 Jan;115(1):37-43. doi: 10.1016/j.clineuro.2012.04.005. Epub 2012 Apr 24. PMID 22537870
- [Background] Stupp R, Mason WP, van den Bent MJ, Weller M, Fisher B, Taphoorn MJ, Belanger K, Brandes AA, Marosi C, Bogdahn U, Curschmann J, Janzer RC, Ludwin SK, Gorlia T, Allgeier A, Lacombe D, Cairncross JG, Eisenhauer E, Mirimanoff RO; European Organisation for Research and Treatment of Cancer Brain Tumor and Radiotherapy Groups; National Cancer Institute of Canada Clinical Trials Group. Radiotherapy plus concomitant and adjuvant temozolomide for glioblastoma. N Engl J Med. 2005 Mar 10;352(10):987-96. doi: 10.1056/NEJMoa043330. PMID 15758009
- [Background] Weller M, Cloughesy T, Perry JR, Wick W. Standards of care for treatment of recurrent glioblastoma--are we there yet? Neuro Oncol. 2013 Jan;15(1):4-27. doi: 10.1093/neuonc/nos273. Epub 2012 Nov 7. PMID 23136223
- [Background] Gempt J, Forschler A, Buchmann N, Pape H, Ryang YM, Krieg SM, Zimmer C, Meyer B, Ringel F. Postoperative ischemic changes following resection of newly diagnosed and recurrent gliomas and their clinical relevance. J Neurosurg. 2013 Apr;118(4):801-8. doi: 10.3171/2012.12.JNS12125. Epub 2013 Feb 1. PMID 23373806
- [Background] Barbagallo GM, Jenkinson MD, Brodbelt AR. 'Recurrent' glioblastoma multiforme, when should we reoperate? Br J Neurosurg. 2008 Jun;22(3):452-5. doi: 10.1080/02688690802182256. PMID 18568742
- [Background] Mandl ES, Dirven CM, Buis DR, Postma TJ, Vandertop WP. Repeated surgery for glioblastoma multiforme: only in combination with other salvage therapy. Surg Neurol. 2008 May;69(5):506-9; discussion 509. doi: 10.1016/j.surneu.2007.03.043. Epub 2008 Feb 8. PMID 18262245
- [Background] Chen MW, Morsy AA, Liang S, Ng WH. Re-do Craniotomy for Recurrent Grade IV Glioblastomas: Impact and Outcomes from the National Neuroscience Institute Singapore. World Neurosurg. 2016 Mar;87:439-45. doi: 10.1016/j.wneu.2015.10.051. Epub 2015 Nov 14. PMID 26585720
- [Background] Hervey-Jumper SL, Berger MS. Reoperation for recurrent high-grade glioma: a current perspective of the literature. Neurosurgery. 2014 Nov;75(5):491-9; discussion 498-9. doi: 10.1227/NEU.0000000000000486. PMID 24991712
- [Background] Franceschi E, Omuro AM, Lassman AB, Demopoulos A, Nolan C, Abrey LE. Salvage temozolomide for prior temozolomide responders. Cancer. 2005 Dec 1;104(11):2473-6. doi: 10.1002/cncr.21564. PMID 16270316
- [Background] Goldman DA, Hovinga K, Reiner AS, Esquenazi Y, Tabar V, Panageas KS. The relationship between repeat resection and overall survival in patients with glioblastoma: a time-dependent analysis. J Neurosurg. 2018 Nov 1;129(5):1231-1239. doi: 10.3171/2017.6.JNS17393. Epub 2018 Jan 5. PMID 29303449
- [Background] Lu VM, Jue TR, McDonald KL, Rovin RA. The Survival Effect of Repeat Surgery at Glioblastoma Recurrence and its Trend: A Systematic Review and Meta-Analysis. World Neurosurg. 2018 Jul;115:453-459.e3. doi: 10.1016/j.wneu.2018.04.016. Epub 2018 Apr 11. PMID 29654958
- [Background] Zhao YH, Wang ZF, Pan ZY, Peus D, Delgado-Fernandez J, Pallud J, Li ZQ. A Meta-Analysis of Survival Outcomes Following Reoperation in Recurrent Glioblastoma: Time to Consider the Timing of Reoperation. Front Neurol. 2019 Mar 26;10:286. doi: 10.3389/fneur.2019.00286. eCollection 2019. PMID 30984099
- [Background] Helseth R, Helseth E, Johannesen TB, Langberg CW, Lote K, Ronning P, Scheie D, Vik A, Meling TR. Overall survival, prognostic factors, and repeated surgery in a consecutive series of 516 patients with glioblastoma multiforme. Acta Neurol Scand. 2010 Sep;122(3):159-67. doi: 10.1111/j.1600-0404.2010.01350.x. Epub 2010 Mar 18. PMID 20298491
- [Background] Raymond J, Darsaut TE, Altman DG. Pragmatic trials can be designed as optimal medical care: principles and methods of care trials. J Clin Epidemiol. 2014 Oct;67(10):1150-6. doi: 10.1016/j.jclinepi.2014.04.010. Epub 2014 Jul 16. PMID 25042688
- [Background] Patel M, Au K, Davis FG, Easaw JC, Mehta V, Broad R, Chow MMC, Hockley A, Kaderali Z, Magro E, Nataraj A, Scholtes F, Chagnon M, Gevry G, Raymond J, Darsaut TE. Clinical Uncertainty and Equipoise in the Management of Recurrent Glioblastoma. Am J Clin Oncol. 2021 Jun 1;44(6):258-263. doi: 10.1097/COC.0000000000000812. PMID 33782334
- [Background] Schucht P. RESURGE: Surgery for recurrent Glioblastoma., https://clinicaltrials.gov/ct2/show/NCT02394626 (2020).
- [Background] Schwartz D, Lellouch J. Explanatory and pragmatic attitudes in therapeutical trials. J Chronic Dis. 1967 Aug;20(8):637-48. doi: 10.1016/0021-9681(67)90041-0. No abstract available. PMID 4860352
- [Background] Raymond J, Darsaut TE, Roy DJ. Recruitment in Clinical Trials: The Use of Zelen's Prerandomization in Recent Neurovascular Studies. World Neurosurg. 2017 Feb;98:403-410. doi: 10.1016/j.wneu.2016.11.052. Epub 2016 Nov 19. PMID 27876665
- [Background] Chaichana KL, Zadnik P, Weingart JD, Olivi A, Gallia GL, Blakeley J, Lim M, Brem H, Quinones-Hinojosa A. Multiple resections for patients with glioblastoma: prolonging survival. J Neurosurg. 2013 Apr;118(4):812-20. doi: 10.3171/2012.9.JNS1277. Epub 2012 Oct 19. PMID 23082884
- [Background] Hoover JM, Nwojo M, Puffer R, Mandrekar J, Meyer FB, Parney IF. Surgical outcomes in recurrent glioma: clinical article. J Neurosurg. 2013 Jun;118(6):1224-31. doi: 10.3171/2013.2.JNS121731. Epub 2013 Mar 15. PMID 23495879
- [Derived] Patel M, Au K, Easaw JC, Davis FG, Young K, Mehta V, Bowden GN, Keough MB, Sankar T, Scholtes F, Chagnon M, L'Esperance G, Yuan Y, Gevry G, Raymond J, Darsaut TE. Repeat resection in recurrent glioblastoma (3rGBM) Trial: A randomized care trial. Neurochirurgie. 2022 Apr;68(3):262-266. doi: 10.1016/j.neuchi.2021.09.001. Epub 2021 Sep 14. PMID 34534565